CLINICAL TRIAL: NCT01478438
Title: A Multicenter "Ablate and Resect" Study of Novilase® Interstitial Laser Therapy for the Ablation of Small Breast Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novian Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-002
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Malignant Tumor
Keywords: Unifocal; 20mm in diameter; measures; 5mm away from the skin and chest
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Treat and Excise (Experimental): All subjects will be treated with Interstitial Laser Therapy (ILT) followed by excision no later than 28 days post ablation.
  Interventions: Device: Novilase Interstitial Laser Therapy

INTERVENTIONS:
Device: Novilase Interstitial Laser Therapy — Image guided Interstitial Laser Ablation of breast tumors
  Other Names: Novilase®

SUMMARY:
This study will determine the rate of complete tumor ablation of small breast cancers (≤ 20mm) by Novilase Interstitial Laser Therapy (ILT), and determine the sensitivity and specificity of imaging (MRI, mammography and ultrasound) in detecting residual tumor post ILT ablation as correlated to histopathology from the post-ablation excision.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 to 80 years of age
* Tumor is well visualized through x-ray mammography or ultrasound imaging and amenable to image guidance therapy (a tumor which is well visualized through imaging can be identified from surrounding breast tissue and does not have margins
* obscured by other structures or artifacts on the images)
* Tumor must be well visualized (as defined above) on MRI
* Definitive pathologic diagnosis by needle core biopsy
* Unifocal malignant tumor that does not exceed 20mm in diameter and measures at least 5mm away from the skin and chest wall
* Cluster of microcalcifications that do not exceed 10 mm in diameter and measures at least 5mm away from the skin and chest wall
* Subjects with or without palpable lymph nodes
* Subjects with mammographic appearance of overall dense parenchymal tissue may be included, as long as a clearly evident marker is present at tumor site
* Subjects with less than 25% intraductal component
* Subject has no clinically significant co-morbidities (i.e. chronic illnesses existing simultaneously with and usually independent of breast cancer) that affect life expectancy. Subject has given written informed consent
* Subject agrees to comply with follow up visits

Exclusion Criteria:

* Subjects younger than 18 years of age
* Pregnant or breast-feeding women
* Tumors poorly visualized by x-ray mammography or ultrasound imaging
* Women who are morbidly obese (>300 lbs)
* Acute or chronic severe renal insufficiency (Glomerular filtration rate (GFR) <30ml/min/1.73 sq.meters)
* Moderate to end-stage kidney disease and a history of severe asthma or allergies
* Tumors measuring greater than 20mm in diameter
* Subjects with advanced stage breast cancer
* Subjects with prior history of cancer in the ILT treated breast
* Subjects with recurrent breast cancer
* Subjects with lobular neoplasm, metastatic carcinoma to breast, sarcoma, Phylloides tumor, or Paget's disease
* Subjects with benign vascular tumor
* Subjects with benign lesions such as fibroadenoma, atypical ductal hyperplasia, sclerosing adenosis, Papilloma, fibrocystic disease of breast
* Subjects with DCIS with microinvasion
* Subjects with a cluster of microcalcifications whose diameter is larger than 10 mm.
* Subjects with extensive intraductal component and other characteristics not well visualized by imaging studies
* Subjects who are BRCA positive.
* Inability to lie prone or supine for one hour
* Currently participating or enrolled in another investigational treatment, device or drug study through follow up
* Undergoing concurrent neoadjuvant therapies for breast cancer
* Cardiac pacemaker or other metallic implants which would prevent patient from safely undergoing MRI scan

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Collect information on the proportion of tumors ablated for sample size calculations in the pivotal trial | one month end point
  Evaluate the rate of complete tumor ablation by Novilase ILT of small breast cancers and characterize the correlation of imaging (MR, US, x-ray) in detecting residual post ablation with histopathology of the excised specimen.
  An individual patient will be considered to have a complete ablation if the pathology results post excision demonstrates that no visible gross residual tumor is present.

SECONDARY OUTCOMES:
To gain experience with the cosmetic outcome and rate of recovery tools | One month end point
  Evaluate satisfaction, utilizing the European Organization for Research and Treatment of Cancer Breast Cancer Specific Quality of Life Questionnaire (EORTC QLQ-BR23) survey and cosmetic outcome utilizing the physician-reported Four-Point Scoring System of Breast Cosmesis.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Schwartzberg, MD, Principal Investigator — Rose Medical Center - Rose Breast Center; Michael Shere, M.D., Principal Investigator — North Bristol NHS Trust: Southmead Hospital - The Breast Care Centre
Locations (12):
- United States (9):
  - The Breast Center of Southern Arizona, Tucson, Arizona
  - Rose Medical Center - Rose Breast Center, Denver, Colorado
  - St. Alexius Breast Care of St. Alexius Medical Center, Bartlett, Illinois
  - Advocate Lutheran General Hospital - Caldwell Breast Center, Park Ridge, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Columbia University Medical Center - Department of Surgery, New York, New York
  - University of Toledo - Eleanor N. Dana Cancer Center Breast Care, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Wheaton Franciscan Health System, Wauwatosa, Wisconsin
- United Kingdom (3):
  - North Bristol NHS Trust: Southmead Hospital - The Breast Care Centre, Bristol
  - Mid Essex Hospital Services NHS Trust: Broomfield Hospital - Breast Unit, Chelmsford
  - Norfolk & Norwich University NHS Foundation Trusts: Norfolk and Norwich University Hospital, Norwich

REFERENCES:
- [Background] Dowlatshahi K, Francescatti DS, Bloom KJ. Laser therapy for small breast cancers. Am J Surg. 2002 Oct;184(4):359-63. doi: 10.1016/s0002-9610(02)00942-x. PMID 12383903
- [Background] Dowlatshahi K, Dieschbourg JJ, Bloom KJ. Laser therapy of breast cancer with 3-year follow-up. Breast J. 2004 May-Jun;10(3):240-3. doi: 10.1111/j.1075-122X.2004.21436.x. PMID 15125752
- See also: Related Info — http://www.novianhealth.com